CLINICAL TRIAL: NCT02379780
Title: Comparison of the Effects of Perioperative Anesthesia Consumption of Ultrasound Guided Subcostal Transversus Abdominis Plane and Paravertebral Block in Laparoscopic Cholecystectomy
Brief Title: Ultrasound Guided Subcostal Transversus Abdominis Plane Versus Paravertebral Block in the Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, specialist dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mengücek gazi hospital
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- USG guided Subcostal TAP block (Active Comparator): after preparing the skin, ultrasound probe was placed obliquely on the upper abdominal wall along the subcostal margin near the midline. the rectus abdominis muscles, transversus abdominis muscles and the fascial plane (TAP) between rectus abdominis and transversus abdominis muscles were identified. after identification, the block needle was introduced anteriorly in the plane of the ultrasound beam. the needle was directed the transversus abdominis plane and 10 ml of bupivacaine (Marcaine 0,25 %) and 5 ml of lidocaine (2%) was injected after negative aspiration.
  Interventions: Procedure: USG guided Subcostal TAP block; Procedure: USG guided Paravertebral Block
- USG guided Paravertebral Block (Active Comparator): prior to start surgery, was performed in the left lateral position. after preparing skin, ultrasound linear probe was placed, 2-3 cm lateral of the T7 / T8 level in the midline. After determining the transverse process and ribs as hyperechoic, the paravertebral space was identified as an area wedge-shaped bounded by the pleura and above the internal intercostal membrane.after identification of the paravertebral space, the block needle was introduced in plane / out of plane and 10 ml of bupivacaine (Marcaine 0,25 %) and 5 ml of lidocaine (2%) was injected after negative aspiration.
  Interventions: Procedure: USG guided Subcostal TAP block; Procedure: USG guided Paravertebral Block

INTERVENTIONS:
Procedure: USG guided Subcostal TAP block — Ultrasonography Assisted Subcostal TAP blockage: In plane technique was applied and 22 G needle (BRAUN Stimuplex D Plus 0,71*50 mm 22G*2) was used. Intravascular injection was eliminated after the passage of rectus sheath by negative aspiration. 0,5-1 ml local anesthetic was applied directly to confirm the right place. 10 cc bupivacain ( 0,5 % Marcain flacon, Astra Zeneca, Sweeden) and 5 cc lidocaine was injected to the site. The same procedure was applied to the opposite site.
  we investigated amount of TIVA during the operation, postoperative Visual Analog Scores and the time that the pain free time.
Procedure: USG guided Paravertebral Block — Ultrasonoraphy assisted Thoracic Paravertebral blockage application: In-plane or out-of-plane technique was used with stimuplex needle (BRAUN Stimuplec D Plus 0,71*50 mm 22 G* 2'', 15°). Popping sensation that was felt by the penetration of the internal intercostal membrane, guided to paravertebral space. Intravascular injection was eliminated by negative aspiration. 0,5 - 1 ml local anesthetic injection was administered to show the displacement of pleura downward that confirmed the place of the needle in the right place. Then 10 cc bupivacain (% 0.5 Marcaine® flacon, Astra Zeneca, Sweeden) and 5 cc lidocaine was injected to the site.
  we investigated amount of TIVA during the operation, postoperative Visual Analog Scores and the time that the pain free time.

SUMMARY:
The investigators aimed to compare the effects of perioperative anesthesia consumption of ultrasound guided subcostal transversus abdominis plane and paravertebral block in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Fifty patients aged 18 - 65 years, American Society of Anesthesiologists (ASA) I-II-III, scheduled for laparoscopic cholecystectomy were enrolled into the study. Patients were allocated into two groups to receive ultrasound guided subcostal transversus abdominis plane block (group T, n=25) or ultrasound guided paravertebral block (group P, n=25). In all patients; anesthesia was induced with iv propofol (2 mg.kg-1) and maintained with total intravenous anesthesia (TIVA) in a mixture of 50 % nitrous oxide and 50 % oxygen with a total gas flow rate of 4 L min-1. Neuromuscular relaxation was induced with iv rocuronium (0.5 mg.kg-1). Propofol (2 mg / cc, 2-4 mg / kg / h) and remifentanil (13.3 mcg / cc, 1-3 mcg / kg / h) combination was used in TIVA. Propofol and remifentanil rates increased or reduced according to the patient's hemodynamic response. Prior to start surgery, ultrasound guided subcostal transversus abdominis plane or paravertebral block was performed in patients .

Blood pressure, heart rate and peripheral oxygen saturation,TIVA consumption of 0, 5, 10, 15, 30, 60 min were recorded for all patients.Before the end of surgery, tramadol was administered (2 mg / kg) for all patients.

All patients were evaluated at postoperative 2th, 4th, 8th, 12th, 24th hours with; operation time, heart rate, blood pressure, peripheral oxygen saturation, visual pain scores (VAS), analgesic consumption, complications (hypotension, anaphylaxis, hematoma, IV injection, intra-abdominal organ injury, pneumothorax ) and patient satisfaction status were recorded. In the postoperative period if there is additional analgesic requirements (VAS≥4) tramadol 2 mg.kg-1 was administered as IV. The first hour is needed analgesia were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years of age,
* ASA I-II-III
* laparoscopic cholecystectomy to be applied

Exclusion Criteria:

* patient refusal
* mental and psychiatric disorders,
* allergy history of the drug to be used,
* kyphoscoliotic anatomical disorder
* patients with coagulopathies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
anesthetic and opioid consumption during operation | six months

SECONDARY OUTCOMES:
postoperative VAS scores | six months
duration of analgesia | six months

CONTACTS AND LOCATIONS:
Overall Officials: ILKE KUPELI, Principal Investigator — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; ZEHRA BEDİR, Study Chair — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; HUSEYIN EKEN, Study Chair — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; UFUK KUYRUKLUYILDIZ, Study Chair — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; DIDEM ONK, Study Chair — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; ORHAN BINICI, Study Chair — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; AYSIN ALAGOL, Study Director — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL; GULDANE KARABAKAN, Study Chair — MENGUCEK GAZI TRAINING AND RESEARCH HOSPİTAL

REFERENCES:
- [Result] Hebbard P. Subcostal transversus abdominis plane block under ultrasound guidance. Anesth Analg. 2008 Feb;106(2):674-5; author reply 675. doi: 10.1213/ane.0b013e318161a88f. No abstract available. PMID 18227342
- [Result] Williams SR, Chouinard P, Arcand G, Harris P, Ruel M, Boudreault D, Girard F. Ultrasound guidance speeds execution and improves the quality of supraclavicular block. Anesth Analg. 2003 Nov;97(5):1518-1523. doi: 10.1213/01.ANE.0000086730.09173.CA. PMID 14570678
- [Result] Cheema SP, Ilsley D, Richardson J, Sabanathan S. A thermographic study of paravertebral analgesia. Anaesthesia. 1995 Feb;50(2):118-21. doi: 10.1111/j.1365-2044.1995.tb15092.x. PMID 7710020
- [Result] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Result] Ozkan D, Akkaya T, Comert A, Balkc N, Ozdemir E, Gumus H, Ergul Z, Kaya O. Paravertebral block in inguinal hernia surgeries: two segments or 4 segments? Reg Anesth Pain Med. 2009 Jul-Aug;34(4):312-5. doi: 10.1097/AAP.0b013e3181ae1169. PMID 19574864
- [Result] Mishriky BM, George RB, Habib AS. Transversus abdominis plane block for analgesia after Cesarean delivery: a systematic review and meta-analysis. Can J Anaesth. 2012 Aug;59(8):766-78. doi: 10.1007/s12630-012-9729-1. Epub 2012 May 24. PMID 22622954
- [Result] Thavaneswaran P, Rudkin GE, Cooter RD, Moyes DG, Perera CL, Maddern GJ. Brief reports: paravertebral block for anesthesia: a systematic review. Anesth Analg. 2010 Jun 1;110(6):1740-4. doi: 10.1213/ANE.0b013e3181da82c8. Epub 2010 May 6. PMID 20448076
- [Result] Aveline C, Le Hetet H, Le Roux A, Vautier P, Cognet F, Vinet E, Tison C, Bonnet F. Comparison between ultrasound-guided transversus abdominis plane and conventional ilioinguinal/iliohypogastric nerve blocks for day-case open inguinal hernia repair. Br J Anaesth. 2011 Mar;106(3):380-6. doi: 10.1093/bja/aeq363. Epub 2010 Dec 21. PMID 21177284